CLINICAL TRIAL: NCT06675227
Title: Comparison of Electrolyte Beverages and Water as Solvents for Bowel Preparation: A Single-Blind, Prospective, Multicenter Randomized Controlled Trial
Brief Title: Comparison of Electrolyte Beverages and Water as Solvents for Bowel Preparation
Acronym: EBSBP-01
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Third Military Medical University (Other)
Collaborators: The thirteenth people's hospital of Chonqing (Unknown); Fuling people's hospital of Chongqing (Unknown)
Responsible Party: Principal Investigator, Weidong Tong, Director, Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20240924; 2022XLC05 (Other Grant/Funding Number: Army Medical University)
Record Dates: First submitted 2024-11-03; First posted 2024-11-05 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Bowel Preparation Before Colonoscopy
Keywords: bowel preparation; Electrolyte Beverages

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drinking Water Group (No Intervention): This group will apply the ordinary drinking water as the solvents for 2L PEG to dissolve.
- Electrolyte Beverages Group (Experimental): This group will apply the electrolyte beverages(Alienergy) instead of ordinary drinking water as the solvents for 2L PEG to dissolve.
  Interventions: Dietary Supplement: electrolyte beverages

INTERVENTIONS:
Dietary Supplement: electrolyte beverages — Using Electrolyte Beverages as replacement for water to dissolve PEG(2L plan) in bowel preparation process.
  Arms: Electrolyte Beverages Group

SUMMARY:
Using Electrolyte Beverages as replacement for water to dissolve PEG(2L plan) in bowel preparation process.

The aim of this study is to test whether Electrolyte Beverages as solvents can improve the cleanness of bowel preparation and the satisfaction of patients.

DETAILED DESCRIPTION:
The application of electronic colonoscopy has shown a significant upward trend in the diagnosis, screening, and health check-ups for colorectal diseases.

To clean the colon, patients must consume several liters of bowel preparation solution in a short period before the procedure.

However, a significant number of patients experience nausea or even vomiting, preventing them from completing the recommended dose, resulting in suboptimal bowel preparation and affecting the colonoscopy process.

Therefore, the investigators have designed a protocol that uses sugar-free electrolyte beverages instead of regular drinking water as a solvent for the laxative solution. By improving the taste of the oral solution and increasing the electrolyte content, the investigators aim to enhance patient compliance with colonoscopy preparation and ultimately assess the effectiveness of bowel cleansing.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy individuals or those with mild or well-controlled chronic diseases.
2. Patients scheduled for outpatient colonoscopy.
3. Patients prescribed sodium phosphate or polyethylene glycol for bowel preparation.
4. Willing to participate and sign the informed consent form.
5. Age ≥18 years
6. ECOG performance status <2

Exclusion Criteria:

1. Patients who refuse to participate in the study.
2. Patients requiring enema preparation.
3. Uncontrolled hypertension.
4. Patients with diabetes.
5. Pregnant patients.
6. Suspected bowel obstruction.
7. Risk of aspiration.
8. Patients with severe ulcerative colitis, gastric retention, bowel perforation, toxic colitis, or megacolon.
9. Patients with severe systemic diseases (including NYHA class 3-4 heart failure, Child-Pugh class C liver failure).
10. Patients with a known allergy to polyethylene glycol.
11. Patients with a history of major gastrointestinal surgery or any other conditions that may interfere with study outcomes or adherence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2766 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The Boston Bowel Preparation Scale | From enrollment to the time point when patients finished colonscopy (within a week).
  The BBPS is a standardized 9-point assessment scale for the colon. The structure of the colon is divided into its three segments: right colon, transverse colon, and left colon. Each segment is classified from 0 to 3 depending on the degree of soiling. The sum total of the three segments represents the degree of soiling, so that a total ≤ 5 points shows poor bowel preparation, while 6-7 shows good bowel preparation, and ≥ 8 very good bowel preparation.

SECONDARY OUTCOMES:
The Palatability | From enrollment to the time point when patients finished colonscopy(within a week).
  The palatability of different bowel preparation regimens will be assessed using a 4-point scale. The scoring system is as follows: 1 = very poor, 2 = poor, 3 = good, 4 = very good. Each participant's score will be collected and statistically analyzed.
Lesion Detection Rate | From enrollment to the time point when patients finished colonscopy (within a week).
  The proportion of polyps, tumors, inflammatory bowel disease, and diverticulosis detected during colonoscopy under different bowel preparation regimens will be recorded. The detection rate will be expressed as a percentage, and differences between the groups will be analyzed.

OTHER OUTCOMES:
Patient Willingness to Repeat | From enrollment to the time point before colonscopy(within a week).
  The willingness of patients to undergo a repeat colonoscopy after the procedure will be recorded and analyzed. This will be quantified using a Yes/No format, and the proportion of willingness in each group will be calculated.
Bowel Preparation Time | From enrollment to the time point before colonscopy(within a week).
  The total time (in minutes) required for each patient to complete 2000 ml of bowel preparation solution will be recorded, and the average time and standard deviation will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Tong, MD, Principal Investigator — Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Locations (1):
- Army Medical Center, Chongqing, Chongqing Municipality, China